CLINICAL TRIAL: NCT01729000
Title: Gloving and Handwashing to Prevent Invasive Infections in Necrotizing Enterocolitis
Brief Title: Study to Determine if Gloving in Addition to Hand Hygiene Will Prevent Invasive Infections and Necrotizing Enterocolitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, David A Kaufman, Prinicpal Investigator, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 13971
Record Dates: First submitted 2011-03-04; First posted 2012-11-20 (Estimated); Last update posted 2012-11-20 (Estimated); Status verified 2012-11

CONDITIONS: Neonatal Infection; Neonatal Necrotizing Enterocolitis
Keywords: prematurity; infection control; necrotizing entercolitis
MeSH Terms: conditions — Enterocolitis, Necrotizing; Premature Birth | interventions — Gloves, Protective

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hand hygiene (No Intervention): All staff that have interaction with subjects will perform hand hygiene with all patient contact and before all contact with the intravenous line.
- Hand hygiene plus gloving (Experimental): All staff that have interaction with subjects will perform hand hygiene and wear gloves with all patient contact and before all contact with the intravenous line.
  Interventions: Other: Gloves

INTERVENTIONS:
Other: Gloves — All staff must wear gloves for subjects that are in the experimental group.
  Arms: Hand hygiene plus gloving

SUMMARY:
The purpose of this study is to compare the additional use of gloves (with handwashing before and after gloving) for all patient contact while infants have intravenous (central or peripheral) access in a RCT. Preterm infants <1000 grams or less than 29 weeks gestational age will be randomized after birth to either a handwashing-gloving group or handwashing only group. The primary outcome will be the incidence of invasive infections (bacterial or fungal) or necrotizing enterocolitis. Secondary outcomes will include hospital days, preterm morbidities, mortality, and hospital costs.

DETAILED DESCRIPTION:
All infants who had a birth weight of less than or equal to 1000 grams or who were born less than 29 weeks gestation were eligible for this study. 120 subjects were randomized by day of life(dol) 8 to one of two study groups--hand hygiene or hand hygiene plus gloving. Study signs were placed at the bedside and on the isolette sides of each infant with the appropriate study group guidelines.

The investigators goal was to target the time period these infants are at high-risk for infection or NEC and its associated mortality. The targeted time was the first 4 weeks of life or longer while intravenous access is still required. The average age for the first episode of late-onset sepsis is 22(+/-0.5) days (median: 17 days; 75th percentile: 28 days; 95th percentile: 57 days). The majority of infections that occur after 4 weeks of life are in patients still requiring IV access (peripheral or central). The presence of an intravenous line in this group of preterm infants correlates with the presence of risk factors for infection that would necessitate the need for intravenous access including: parenteral nutrition, lipid infusion, use of broad spectrum antibiotics, and the intravenous line itself (if it is a central venous catheter). This strategy focused on the individual infant's risks, limits exposure to and decreases cost of intervention.

ELIGIBILITY:
Inclusion Criteria:

* Birth weight <1000 grams or gestational age ≤28 weeks
* less than or equal to 7 days of age

Exclusion Criteria:

* greater than 7 days of age

Max Age: 8 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 124 (Actual)
Dates: Start 2008-10; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Invasive Infection | Participants will be followed during their NICU hospitalization, an expected average of 3 months
  Invasive infection will be defined as growth of bacteria from culture (blood, urine, CSF, peritoneal) with clinical signs and symptoms of sepsis
Necrotizing enterocolitis (NEC) | Participants will be followed for their entire NICU hospitalization, which is an average of 3 months
  NEC will be defined as stage II or greater using Bell's modified criteria

SECONDARY OUTCOMES:
Length of stay | Participants will be followed for their entire NICU hospitalization, which is an average of 3 months
  Length of stay will be compared in each study arm
Mortality | Participants will be followed for their entire NICU hospitalization, which is an average of 3 months
  Mortality will be compared in each study arm
Hospital cost | Participants will be followed for their entire NICU hospitalization, which is an average of 3 months
  Hospital costs will be compared in each study arm
Common neonatal morbidities | Participants will be followed for their entire NICU hospitalization, which is an average of 3 months
  Common morbidities will be compared in each study arm

CONTACTS AND LOCATIONS:
Overall Officials: David A Kaufman, MD, Principal Investigator — University of Virginia School of Medicine
Locations (1):
- University of Virginia, Newborn Intensive Care Unit, Charlottesville, Virginia, United States

REFERENCES:
- [Derived] Kaufman DA, Blackman A, Conaway MR, Sinkin RA. Nonsterile glove use in addition to hand hygiene to prevent late-onset infection in preterm infants: randomized clinical trial. JAMA Pediatr. 2014 Oct;168(10):909-16. doi: 10.1001/jamapediatrics.2014.953. PMID 25111196